CLINICAL TRIAL: NCT05529147
Title: The Effects of Medication Induced Blood Pressure Reduction on Cerebral Hemodynamics in Hypertensive Frail Elderly
Acronym: BLUEBERRY
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL80929.091.22; 2022-001283-10 (EudraCT Number)
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2022-08

CONDITIONS: Hypertension; Frailty; Old Age; Dementia; Orthostatic Intolerance; Orthostatic Hypotension; Cerebral Hypoperfusion
MeSH Terms: conditions — Hypertension; Frailty; Alzheimer Disease; Orthostatic Intolerance; Hypotension, Orthostatic | interventions — Antihypertensive Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antihypertensive Agents — Study participants receive antihypertensive drug treatment as part of regular care to induce systolic BP (SBP) reductions ≥10 mmHg within 6-8 weeks, while reaching a treatment target of ≤140 mmHg, and while preserving diastolic BP ≥70 mmHg.

SUMMARY:
Rationale: Systolic hypertension represents the leading risk for burden of disease among older adults (age >70 years), with an increasing prevalence due to the increase in lifespan. Antihypertensive drug treatment (AHT) is beneficial in fit (non-frail) older adults, with substantial (≈40 %) risk reductions for cardiovascular events and mortality. Scarce evidence exists on the risks of adverse effects related to AHT. It has been suggested in medical literature that AHT in frail elderly might cause cerebral hypoperfusion and/or orthostatic hypotension. Therefore, current guidelines advise clinicians to be more cautious regarding treatment targets in this population. However, the evidence for these adverse effects is limited to observational and cross-sectional data and opinion pieces. In contrast to the suggestion of potential adverse effects of AHT in elderly, recent experimental data and secondary analyses of clinical trials do not provide support for this statement. However, evidence in frail older patients remains scarce. Studies that directly examine the safety of AHT with regard to cerebral hemodynamics and orthostatic tolerance in frail elderly are needed to inform potential changes in current treatment guidelines and prevent undertreatment of hypertension in frail older patients.

Objective: To examine the impact of medication induced systolic BP (SBP) reductions ≥10 mmHg, while reaching a treatment target of ≤140 mmHg, on cerebral blood flow (CBF) in frail elderly with untreated or uncontrolled systolic hypertension at baseline. We hypothesise that these blood pressure lowering targets (which are consistent with clinical guidelines for non-frail older patients) are not accompanied by detrimental reductions in CBF (i.e. >10% from baseline).

Study design: An explorative observational study will be performed to examine the effects of medication induced SBP reductions ≥10 mmHg to office SBP ≤140 mmHg on CBF in frail elderly with untreated or uncontrolled hypertension. Participants will be treated as in usual patient care for older adults with hypertension. Participants will undergo one baseline assessment before exposure to (additional) AHT, followed by in duplo follow-up assessments 6-10 weeks after the start of AHT. The in duplo follow-up evaluations will be performed on separate days within 2 weeks while continuing treatment.

Study population: Twelve frail (Clinical Frailty Scale 4-7) elderly (age ≥70 years) with untreated or uncontrolled systolic hypertension (office SBP ≥150 mmHg) that will be subjected to (additional) AHT as part of regular care.

Main study parameters/endpoints: The change in resting CBF from baseline to follow-up (i.e. the average of the in duplo follow-up assessments). Secondary outcomes relate to cerebrovascular autoregulation (CA) and orthostatic tolerance.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects will be subjected to AHT, essentially identical to what is considered 'guideline care', while their wellbeing will be monitored closely. Since all study procedures and used measurement techniques are non-invasive, the nature and extent of burden and risks associated with participation and measurements are negligible.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years.
* Clinical Frailty Scale ≥4 and ≤7.
* Diagnosis of:

  * Untreated systolic hypertension, i.e. unattended office SBP ≥150 mmHg without AHT, or;
  * Uncontrolled systolic hypertension, i.e. unattended office SBP ≥150 mmHg despite AHT.
* Will be starting (untreated) or adding (uncontrolled) AHT in the near future for (further) reducing SBP by ≥10 mmHg while reaching a treatment target of unattended office SBP

  ≤140 mmHg, while keeping unattended office diastolic blood pressure ≥70 mmHg, with the indication of primary or secondary prevention of vascular events, judged by the treating physician (geriatrician or primary care physician)
* Able to understand and perform study related procedures.

Exclusion Criteria:

* Unable to provide signed and dated informed consent form.
* Mentally incompetent subjects (e.g. due to dementia) as assessed by a physician.
* Currently enrolled in another interventional study targeting either BP and/or CBF.
* Cardiovascular event within the past 3 months.
* Estimated glomerular filtration rate (eGFR) <40 ml/min.
* Known secondary cause of hypertension that causes safety concerns.

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Hypertensive frail older adults
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Change in MCAv across follow-up | 6-8 weeks
  The primary study parameter is the relative change in CBF from baseline to follow-up (i.e. the average of the in duplo follow-up assessments), measured as the mean bilateral CBF velocity in the MCA (in cm/s).

SECONDARY OUTCOMES:
Changes in cerebral autoregulation and orthostatic tolerance | 6-8 weeks
  The relative and absolute changes in measures of CA (i.e. dCA and BRS) and OT from baseline to follow-up. Regarding OT, it will also be evaluated whether the incidence of orthostatic hypotension differs between baseline and follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen A Claassen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weijs RWJ, de Roos BM, Thijssen DHJ, Claassen JAHR. Intensive antihypertensive treatment does not lower cerebral blood flow or cause orthostatic hypotension in frail older adults. Geroscience. 2024 Oct;46(5):4635-4646. doi: 10.1007/s11357-024-01174-4. Epub 2024 May 9. PMID 38724874